CLINICAL TRIAL: NCT02220478
Title: A Prospective Controlled Study on Signature Anterior Posterior/Lateral Acetabular Cup Placement System in Total Hip Arthroplasty
Brief Title: Signature Acetabular Posterior/Lateral Data Collection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to engage surgeons to participate in the study
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO.CR.GH24
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Noninflammatory Degenerative Joint Disease; Avascular Necrosis; Rheumatoid Arthritis
Keywords: hip; Signature
MeSH Terms: conditions — Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Signature Cutting Guides (Active Comparator): Patients indicated for a Posterior Lateral THA utilizing non implantable Signature Cutting Guides during surgery.
  Interventions: Device: Posterior Lateral Approach Total Hip Arthroplasty
- Conventional Instrumentation (Active Comparator): Patients indicated for a Posterior Lateral THA utilizing non implantable Conventional Instrumentation during surgery.
  Interventions: Device: Posterior Lateral Approach Total Hip Arthroplasty

INTERVENTIONS:
Device: Posterior Lateral Approach Total Hip Arthroplasty — All patients enrolled in the study are indicated for a total hip replacement, and will receive this replacement from the surgeon via a Posterior Lateral surgical approach.

SUMMARY:
The primary purpose of this pilot study is to evaluate the accuracy of cup placement between two instrumentation technologies: Cutting Guide and Conventional Instrumentation.

DETAILED DESCRIPTION:
Using a more advanced surgical technique may assist surgeons and patients in a variety of ways including identifying a specific-size for the prosthesis prior to surgery, increasing operating room efficiency, and reducing the number of traditional instruments needed. This may reduce cost associated with the instrument inventory and instrument sterilization. Operating time may also be reduced, potentially decreasing the patient's risk of infection. However, before these hypotheses can be tested, it is important to fully understand the efficacy and accuracy of Signature Custom Guides and their use in Total Hip Arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with one of the following indication:
* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Rheumatoid arthritis.
* Correction of functional deformity.
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques.

Additional inclusion criteria include:

* Subjects requiring primary total hip arthroplasty
* 20 to 75 years of age
* Subjects with a diagnosis of osteoarthritis or traumatic arthritis
* Subjects willing to return for follow-up evaluations.
* Subjects who can read, understand study information and give written consent without representation of a legally authorized representative.
* Bilateral patients are included if staged.
* Only Posterior Lateral Approach can be used for inclusion in this study

Exclusion Criteria:

- Exclusion criteria should be in accordance with Contraindications for the Biomet primary acetabular cup.

Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement.

Additional contraindications include:

* Subjects whose bony structure deviates substantially from the general norm sufficiently to require non-standard implants. Specific examples of these are total dislocation of the hip, severe coxa vera deformity, and severe forms of multiple epiphyseal dysplasia
* Subjects unable to cooperate with and complete the study
* Dementia and inability to understand and follow instructions
* Neurological conditions affecting movement
* Pregnancy

Additional exclusion criteria include:

* Surgical approach other than posterior lateral.
* Simultaneous bilateral procedures

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, Ph.D., Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Signature Cutting Guides | Conventional Instrumentation
Started | 14 | 10
Completed | 11 | 9
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Signature Cutting Guides | Conventional Instrumentation | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.9) | 68.8 (6.4) | 62.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 0 | 11
  France | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Operative Room Time
Description: Average operative time
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Signature Cutting Guides | Conventional Instrumentation
Number analyzed (Participants) | 14 | 10
minutes | 84.7 (12.0) | 78.3 (3.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Signature Cutting Guides | Conventional Instrumentation
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 1/14 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Signature Cutting Guides (N=14) | Conventional Instrumentation (N=10)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No